CLINICAL TRIAL: NCT01293968
Title: Therapeutic Effects of "Ibuprofen, Diphenhydramine and Aluminium MgS" on Recurrent Aphthous Stomatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pantea Nazeman, Miss, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: qums353
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-05

CONDITIONS: Aphthous Stomatitis
Keywords: Aphthous Stomatitis; Ibuprofen; treatment efficacy
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — Ibuprofen; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5cc Ibuprofen100mg,10 cc Diphenhydramine25mg,10 cc AlMgS550mg (Experimental)
  Interventions: Drug: Ibuprofen, Diphenhydramine and Aluminium MgS
- 100 cc Diphenhydramine, 25 mg and 100 cc AlMgS 550 mg (Active Comparator)
  Interventions: Drug: Diphenhydramine and Aluminium MgS

INTERVENTIONS:
Drug: Ibuprofen, Diphenhydramine and Aluminium MgS — 3 times daily for 3 days
  Arms: 5cc Ibuprofen100mg,10 cc Diphenhydramine25mg,10 cc AlMgS550mg
Drug: Diphenhydramine and Aluminium MgS — 3 times daily for 3 days
  Arms: 100 cc Diphenhydramine, 25 mg and 100 cc AlMgS 550 mg

SUMMARY:
The intention of the study is to study the effects of Ibuprofen, Diphenhydramine and Aluminium MgS in decreasing the signs of recurrent aphthous stomatitis (RAS)

DETAILED DESCRIPTION:
Recurrent aphthous stomatitis (RAS) is the most painful oral lesion with a considerable prevalence . The most common aphthous ulcer treatments include applying topical agents such as antibiotics, Non Steroidal Anti Inflammatory Drugs (NSAIDs) to immunosuppressants.

The mixture of Diphenhydramine and Aluminum MgS suspension has been prescribed as an analgesic mouthwash for a long time in order to decrease a great number of oral ulcers symptoms such as aphthous ulcers. Ibuprofen is a potent NSAID with fair anti-inflammatory potential prescribed in dental pains.

This double-blind randomized clinical trial was conducted to assess the effect of Ibuprofen, Diphenhydramine and Aluminium MgS mixture on symptoms of aphthous ulcers.40 patients will be participating in this study,20 will receive the mixture of Diphenhydramine and Aluminium MgS while the other group will receive Ibuprofen, Diphenhydramine and Aluminium MgS mixture.

All patients will be instructed to apply the drug on the site of the ulcer 30-60 minutes before meals, 3 times daily. The ulcers will be assessed when the drug is applied for 3 days and the level of pain and irritation will be estimated by VAS (Visual Analogue Scale, a scaled ruler which the zero point displays the zone of lack of pain and the 10th point was considered as the zone of maximum pain).

ELIGIBILITY:
Inclusion Criteria:

* possessing at least one painful aphthous ulcer in the last 3 days
* older than 10 years of age

Exclusion Criteria:

* systemic disease or specific syndrome (such as Behcet's)
* pregnancy
* breastfeeding
* allergy to NSAIDs
* history of asthma, peptic ulcers, hepatic and renal failures and hemorrhagic disorders
* consumption of anti-inflammatory medications in the last 24 hours

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katayun Borhanmojabi, D.D.S,M.S, Study Chair — QUMS; Katayun Borhanmojabi, D.D.S,M.S, Study Director — QUMS; Marjan Nasiri asl, PhD, Study Director — QUMS; Faeze Mirmiran, D.D.S, Principal Investigator — QUMS; Pantea Nazeman, student, Principal Investigator — QUMS
Locations (2):
- Iran (2):
  - Dental faculty of Qazvin University of Medical Sciences, Qazvin, Qazvin Province
  - Qazvin University of Medical sciences, Qazvin, Qazvin Province

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibuprofen, Diphenhydramine and Aluminium MgS | Diphenhydramine and Aluminium MgS
Started | 20 | 17
Completed | 17 | 14
Not Completed | 3 | 3
Not completed — non-cooperation | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen, Diphenhydramine and Aluminium MgS | Diphenhydramine and Aluminium MgS | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 16 | 13 | 29
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.4 (10.04) | 32.0 (10.0) | 32.2 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Effect of Ibuprofen, Diphenhydramine and Aluminium MgS Measured on Decrease in Pain Level and Burning Sensation
Description: pain sensation was measured by VAS (Visual Analogue Scale, a scaled ruler which the zero point displays the zone of lack of pain and the 10th point was considered as the zone of maximum pain)) 4 days after the consumption of the solution
Time Frame: four days after the start of the study
Population: The intention of the study is to study the effects of Ibuprofen, Diphenhydramine and Aluminium MgS in decreasing the signs of RAS
Measure: Mean (95% Confidence Interval); unit: scores in Visual Analogue Scale
Groups:
- Ibuprofen, Diphenhydramine and Aluminium MgS: the group received the study solution containing 5cc ibuprofen 100mg, 10 cc Diphenhydramine 25 mg and 10 cc AlMgS which was applied on the ulcers 30-60 minutes before meals, 3 times daily for 3 days
- Diphenhydramine and Aluminium MgS: the group received the placebo solution containing 10 cc Diphenhydramine 25 mg and 10 cc AlMgS which was applied on the ulcers 30-60 minutes before meals, 3 times daily for 3 days
Arm/Group | Ibuprofen, Diphenhydramine and Aluminium MgS | Diphenhydramine and Aluminium MgS
Number analyzed (Participants) | 17 | 14
scores in Visual Analogue Scale | 3.176 [1.169 to 5.183] | 3.821 [2.028 to 5.614]

2. Secondary Outcome: The Effect of Ibuprofen, Diphenhydramine, Aluminium MgS and Diphenhydramine and Aluminium MgS in Decreasing the Pain Level and Burning Sensation
Description: pain sensation was measured by VAS (Visual Analogue Scale) 4 days after the consumption of the solutions and the results of both drugs was analyzed
Time Frame: 4 days after the solution consumption
Reporting Status: Not Posted
Measure: unit: scales in Visual Analogue Scale

ADVERSE EVENTS:
Arm/Group | Ibuprofen, Diphenhydramine and Aluminium MgS | Diphenhydramine and Aluminium MgS
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14

LIMITATIONS AND CAVEATS:
Small number of population. Studying just one concentration of Ibuprofen. Lack of a placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes